CLINICAL TRIAL: NCT07121205
Title: Comparative Analysis of High-Dose Dual Therapies in First-Line Helicobacter Pylori Eradication: A Multicenter Retrospective Study
Brief Title: High-Dose Dual Therapy for H. Pylori Eradication (RETRO-HP Study)
Acronym: RETROHP
Status: Completed | Type: Observational
Sponsor: Liyueyue (Other)
Collaborators: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor-Investigator, Liyueyue, Associate Professor, Qilu Hospital of Shandong University
Organization: Qilu Hospital of Shandong University (Other)
Other Study IDs: KYLL-2025-07-009; KYLL-2025-07-009 (Other: Qilu Hospital of Shandong University)
Record Dates: First submitted 2025-08-04; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: HELICOBACTER PYLORI INFECTIONS
Keywords: Helicobacter pylori; dual therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — De-identified clinical data from medical records (e.g., treatment history, adverse events) were stored in encrypted Excel files. No biological samples retained.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- VA-10 day group
  Interventions: Other: This study is a retrospective study, and all data have been collected in advance with no active intervention required.
- VA-14 day group
  Interventions: Other: This study is a retrospective study, and all data have been collected in advance with no active intervention required.
- TA group
  Interventions: Other: This study is a retrospective study, and all data have been collected in advance with no active intervention required.
- EA group
  Interventions: Other: This study is a retrospective study, and all data have been collected in advance with no active intervention required.

INTERVENTIONS:
Other: This study is a retrospective study, and all data have been collected in advance with no active intervention required. — This study is a retrospective study, and all data have been collected in advance with no active intervention required.

SUMMARY:
Background:

High-dose dual therapy (HDDT) has emerged as a potential first-line treatment for Helicobacter pylori infection, but its efficacy and safety across different regimens and populations remain unclear. This study aimed to compare real-world outcomes of various HDDT protocols and identify factors influencing treatment failure.

Methods:

A multicenter retrospective analysis was conducted using data from 15 medical centers (January 2022-January 2025). Patients received one of four HDDT regimens: vonoprazan-amoxicillin for 10 days (VA-10) or 14 days (VA-14), esomeprazole-amoxicillin (EA), or tegoprazan-amoxicillin (TA). Primary outcomes included eradication rates (modified intention-to-treat analysis) and adverse events.

DETAILED DESCRIPTION:
This study is a multicenter, retrospective, observational study utilizing medical records of outpatients who received standard high-dose dual therapy (HDDT) for Helicobacter pylori eradication between January 2022 and January 2025. The aim was to compare the efficacy and adverse event rates of different HDDT regimens.

Collected data included:

Baseline demographics (age, sex, etc.)

Medical/lifestyle history

Treatment regimens

Adverse events

Compliance

All data were anonymized at collection, and no additional patient contact or information collection was required. Since this study involved only retrospective chart review without new interventions, patient consent was waived by the ethics committee.

Treatment Groups

Patients were categorized based on their actual prescribed regimens:

Amoxicillin + Vonoprazan (10-day course)

Amoxicillin + Vonoprazan (14-day course)

Amoxicillin + Tegoprazan (14-day course)

Amoxicillin + Esomeprazole (14-day course)

These groups were compared to assess differences in H. pylori eradication rates.

Study Characteristics No active intervention or real-time questionnaire collection was involved.

Complies with the real-world evidence (RWE) framework for retrospective studies.

Primary Outcome Eradication rate comparison between HDDT regimens (assessed via modified intention-to-treat analysis).

Secondary Outcomes Adverse event rates across different HDDT regimens.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients aged 18-70 years, regardless of gender; (2) absent history of receiving H. pylori eradication therapy; (3) diagnosed with H. pylori infection through at least one of the following methods: rapid urease test, ¹³C/¹⁴C-urea breath test, or histopathological examination.

Exclusion Criteria:

* (1) patients with incomplete medical records, including missing treatment details, absence of post-treatment follow-up test results, or failure to complete essential follow-up assessments; (2) patients who received treatment regimens that did not conform to the standardized HDDT protocol specified in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (1) patients aged 18-70 years, regardless of gender; (2) absent history of receiving H. pylori eradication therapy; (3) diagnosed with H. pylori infection through at least one of the following methods: rapid urease test, ¹³C/¹⁴C-urea breath test, or histopathological examination.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Eradication rate | 4-6 weeks
  Comparison of Eradication Rates among Four Different High-Dose Dual Therapies for Helicobacter pylori
Comparison of Eradication Rates Among Four Different High-Dose Dual Therapies for Helicobacter pylori | 4-6 weeks

SECONDARY OUTCOMES:
Adverse Events and Compliance | 4-6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Qilu Hospital of Shandong University, Jinan, Shandong, China., Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wiklund AK, Santoni G, Yan J, Radkiewicz C, Xie S, Birgisson H, Ness-Jensen E, von Euler-Chelpin M, Kauppila JH, Lagergren J. Risk of Gastric Adenocarcinoma After Eradication of Helicobacter pylori. Gastroenterology. 2025 Aug;169(2):244-250.e1. doi: 10.1053/j.gastro.2025.01.239. Epub 2025 Feb 7. PMID 39924057
- [Background] Park JY, Georges D, Alberts CJ, Bray F, Clifford G, Baussano I. Global lifetime estimates of expected and preventable gastric cancers across 185 countries. Nat Med. 2025 Sep;31(9):3020-3027. doi: 10.1038/s41591-025-03793-6. Epub 2025 Jul 7. PMID 40624406